CLINICAL TRIAL: NCT04926649
Title: The High-frequency Low-volume Ventilation (HFLVV) for Hypoxemia During the Weaning From Cardiopulmonary Bypass in Robot-assisted Cardiac Surgery
Brief Title: HFLVV for Hypoxemia in Robot-assisted Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Qingxiang Mao, Professor, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-59
Record Dates: First submitted 2021-05-31; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Hypoxemia
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional ventilation group (Sham Comparator): Conventional SLV and complementary with DLV when necessary. When SLV was initiated, the patient was ventilated with left lung. FiO2 of 1.0, tidal volume of 6ml/kg, respiratory rate of 16-24 bpm, PEEP of 5-10 cmH2O. The right lung was totally collapsed. If the SpO2 decreased lower than 90%, DLV was started and the operation was paused until the SpO2 increased to 100%. Then the operation was restarted.
  Interventions: Procedure: Differential ventilation to the non-dependent lung
- CPAP group (Active Comparator): SLV of left lung and CPAP of right lung, and complementary with DLV when necessary.
  When SLV was initiated, the patient was ventilated with left lung. FiO2 of 1.0, tidal volume of 6ml/kg, respiratory rate of 16-24 bpm, PEEP of 5-10 cmH2O. After the right lung was totally collapsed, CPAP was started with the pressure less than 8 cmH2O. If SpO2 decreased lower than 90%, DLV was started and the operation was paused until the SpO2 increased to 100%. Then the operation was restarted.
  Interventions: Procedure: Differential ventilation to the non-dependent lung
- HFLVV group (Experimental): SLV of left lung and HFLVV of right lung, and complementary with DLV when necessary.
  When SLV was initiated, the patient was ventilated with left lung. FiO2 of 1.0, tidal volume of 6ml/kg, respiratory rate of 16-24 bpm, PEEP of 5-10 cmH2O. After the right lung was totally collapsed, HFLVV was started with tidal volume of 2ml/kg, respiratory rate of 60 bpm. If SpO2 decreased lower than 90%, DLV was started and the operation was paused until the SpO2 increased to 100%. Then the operation was restarted.
  Interventions: Procedure: Differential ventilation to the non-dependent lung

INTERVENTIONS:
Procedure: Differential ventilation to the non-dependent lung — When the hypoxemia occurs during sing lung ventilation in robot-assisted cardiac surgery, the non-dependent lung will be ventilated with normal tidal volume in conventional ways and the surgery procedure have to be ceased. In this trial, the non-dependent lung will be ventilated with the continuous positive airway pressure (CPAP) or the high-frequency low-volume ventilation (HFLVV) to prevent the hypoxemia.

SUMMARY:
These robot-assisted cardiac surgeries usually require single-lung ventilation (SLV) to facilitate surgical exposure. SLV creates ventilation/perfusion mismatch and shunt (Qs:Qt) through the collapsed lung and leads to hypoxemia. Pulmonary gas exchange often deteriorates after cardiopulmonary bypass (CPB) because of ischemic tissue damage. In some cases, severe hypoxemia may require the cessation of surgical procedures and the initiation of double-lung ventilation to improve oxygenation. In this study, the investigator applied the continuous positive airway pressure (CPAP) or the high-frequency low-volume ventilation (HFLVV) to the non-dependent lung (differential ventilation) during the weaning from CPB. The investigator hypothesized that the differential ventilation would produce the least interference with the surgeon's exposure and better oxygenation. The investigators evaluate the airway pressure, shunt fraction, PaO2/FiO2, cerebral oximetry, surgical field condition and the length of stay in intensive care unit of patients underwent the robot-assisted cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for robot-assisted cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* age <18 or > 70 years
* PaO2/FiO2 ratio < 300 mmHg before anesthesia induction
* American Society of Anesthesiologist (ASA) Grade > 3
* Patients who were converted to conventional open-chest procedure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2022-03-15 (Estimated)

PRIMARY OUTCOMES:
Changes of arterial PaO2 | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Arterial PaO2 (in mmHg) defined as a measurement of partial pressure of oxygen in arterial blood
Changes of PaO2/FiO2 ratio | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  PaO2/FiO2 ratio defined as the ratio of PaO2 to fractional inspired oxygen (FiO2 expressed as a fraction)

SECONDARY OUTCOMES:
Changes of Heart rate | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV
  Heart rate in beat per minute
Changes of mean blood pressure | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  mean blood pressure in mmHg
Changes of cardiac stroke volume variation | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Cardiac stroke volume variation in percentages
Changes of venous pressure of jugular vein | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Venous pressure of jugular vein in cmH2O
Changes of tidal volume | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Tidal volume of both lungs in milliliter
Changes of respiratory rates | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Respiratory rates of both lungs in breath per minute
Changes of airway pressure | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Airway pressure of both lungs in mmHg
Changes of end-tidal carbon dioxide tension | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  End-tidal carbon dioxide tension in mmHg
Changes of blood oxygen saturation | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Blood oxygen saturation of both upper and lower extremities in percentages
Changes of the pulmonary shunt fraction | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  Qs/Qt = ((CcO2 - CaO2) / (CcO2 - CvO2)) * 100
Changes of regional cerebral oxygen saturation | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  regional cerebral oxygen saturation in percentages
Changes of the surgical field | 5 min after induction of anesthesia during DLV, 5 min after SLV, 5 min after HFLVV, 5 min after CPB flow reduced to 1/3, 5min after CPB flow reduced to 2/3, 15min after resuming of DLV]
  The surgeon's evaluation of the surgical field, graded from 0 (no interference) to 3 (maximal interference)

CONTACTS AND LOCATIONS:
Overall Officials: Qingxiang Mao, M.D., Ph.D., Principal Investigator — Daping Hospital, Army Medical University
Locations (1):
- Daping Hospital, Army Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kremer R, Aboud W, Haberfeld O, Armali M, Barak M. Differential lung ventilation for increased oxygenation during one lung ventilation for video assisted lung surgery. J Cardiothorac Surg. 2019 May 6;14(1):89. doi: 10.1186/s13019-019-0910-2. PMID 31060627